CLINICAL TRIAL: NCT04013256
Title: Controlled Human Exposure and THS Generation Core
Brief Title: Controlled Exposure of Healthy Nonsmokers to Secondhand and Thirdhand Cigarette Smoke
Acronym: THS04
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: The human exposure facility was closed by the University.
Sponsor: University of California, San Francisco (Other)
Collaborators: Tobacco Related Disease Research Program (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 28PT-0081
Record Dates: First submitted 2019-06-25; First posted 2019-07-09 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Pollution; Exposure; Smoke Inhalation; Exposure to Pollution
MeSH Terms: conditions — Smoke Inhalation Injury

STUDY DESIGN:
Intervention Model Description: Crossover assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dermal Exposure to Thirdhand Cigarette Smoke (Experimental): Participants will wear clothing that has been exposed to cigarette smoke, for 3 hours while breathing filtered, temperature and humidity controlled air.
  Interventions: Other: Cigarette Smoke
- Inhalational Exposure to Thirdhand Cigarette Smoke (Active Comparator): Participants will breathe cigarette smoke aerosol that has been aged for 22 hours, for 3 hours while wearing clean clothing.
  Interventions: Other: Cigarette Smoke
- Inhalational Exposure to Secondhand Cigarette Smoke (Active Comparator): Participants will breathe cigarette smoke aerosol that has been aged for 30 minutes, for 3 hours while wearing clean clothing.
  Interventions: Other: Cigarette Smoke
- Clean Air Exposure (Sham Comparator): Participants will breathe filtered, temperature and humidity controlled air while wearing clean clothing for 3 hours.
  Interventions: Other: Clean Air and Clean Clothing/Sham exposure

INTERVENTIONS:
Other: Cigarette Smoke — Cigarette smoke, generated by a smoking machine and aged is used to reproduce exposure to secondhand and thirdhand cigarette smoke.
  Arms: Dermal Exposure to Thirdhand Cigarette Smoke; Inhalational Exposure to Secondhand Cigarette Smoke; Inhalational Exposure to Thirdhand Cigarette Smoke
Other: Clean Air and Clean Clothing/Sham exposure — Clean air, created by high-efficiency particulate air (HEPA) and charcoal filtration and temperature and humidity control.
  Clean cotton clothing.
  Arms: Clean Air Exposure

SUMMARY:
This study compares the health effects of dermal and inhalational exposure to thirdhand cigarette smoke to those of inhalational exposure to secondhand cigarette smoke in healthy, adult nonsmokers. Our hypothesis is that dermal exposure increases exposure to the tobacco specific carcinogen, NNK and may affect both endothelial function and epidermal integrity.

DETAILED DESCRIPTION:
Thirdhand cigarette smoke is the smoke chemicals that persist in the environment after smoking. Indoors, they can be found both on surfaces and in the air. Thirdhand smoke derives from secondhand smoke and contains the chemicals that stick to surfaces, are re-emitted into the air and that form by chemical reactions both on surfaces and in the air.

Thirdhand smoke can contain higher concentrations of the tobacco-specific nitrosamine and known carcinogen 4-(methylnitrosamino)-1-(3-pyridyl)-1-butanone (NNK) than secondhand smoke, because nicotine reacts to form NNK in the indoor environment. Dermal exposure to thirdhand smoke includes nicotine, NNK and other tobacco-specific nitrosamines, polycyclic aromatic hydrocarbons, and volatile organic compounds. Inhalational exposure to thirdhand smoke includes nicotine, ultrafine particles and volatile organic compounds. Previous studies have shown that inhalational exposure to secondhand cigarette smoke causes endothelial dysfunction, which is a risk factor for heart disease and heart attacks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy on the basis of medical history, blood pressure and test of C-reactive protein, lipids and blood sugar.
* Non-smoker not exposed to second-hand smoke (SHS) as determined by saliva cotinine < 10 ng/ml and tetrahydrocannabinol (THC) < 50 ng/ml.
* Flow mediated dilation of 4% or greater at screening visit.

Exclusion Criteria:

* Age 18 < or > 50 Physician diagnosis of asthma, heart disease, hypertension, thyroid disease, diabetes, renal or liver impairment or glaucoma.

Unstable psychiatric condition (such as current major depression, history of schizophrenia or bipolar disorder) or current use of more than two psychiatric medications Systolic blood pressure > 150 Diastolic blood pressure > 100 Blood glucose > 110 LDL >130 Pregnancy or breastfeeding (by urine Human Chorionic Gonadotropin (hCG) and/or history) Alcohol or illicit drug dependence within the past 5 years BMI > 35 and < 18 Current illicit drug use (by history or urine test) More than 1 pack year smoking history Ever a daily marijuana smoker Smoked anything within the last 3 months Unable to hold allergy or other over-the-counter (OTC) medicines Occupational exposure to smoke, dusts and fumes Concurrent participation in another clinical trial Unable to communicate in English No social security number

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2020-01-20 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Changes in flow-mediated dilation (FMD) of the brachial artery, caused by pollution exposures, measured by ultrasound | Baseline (before exposure) 30 minutes (after 30 minutes exposure) and 3 hours.
  High-resolution ultrasound of right brachial artery is performed 1 cm distal to antecubital fossa with a 10 megahertz (MHz) linear array probe coupled to a General Electric (GE) Vivid 7 Imaging System. To assess endothelium-dependent dilation, after recording baseline B-mode ultrasound images of the brachial artery and spectral Doppler images of flow velocity, a forearm cuff is inflated to 250 mmHg for 5 minutes to induce reactive hyperemia. Immediately after deflation, Doppler images are obtained to measure reactive hyperemia. FMD of brachial artery will be determined every 15 seconds between 30 and 120 seconds after cuff deflation to capture maximal dilation.The % FMD will be calculated as ratio between the maximum post cuff release brachial artery diameter and baseline diameter. By comparing changes in FMD before exposure, after exposure and next day, we will be able to assess effects of exposure on endothelial function and the potential recovery from these effects.

SECONDARY OUTCOMES:
Changes in trans-epidermal water loss caused by pollution exposures, comparing intact skin to tape-stripped skin | Baseline, 30 minutes, 3 hours, 2 days, 5 days
  We will measure trans-epidermal water loss (TEWL) on the volar forearm using a dermal relative humidity monitor (model IP52, Delfin Technologies Inc.) on adjacent circles of intact skin and skin that has been tape stripped prior to exposure. By comparing changes in TEWL at these two sites, before and after exposure and at day 2 and day 5, we will be able to detect any effects of dermal cigarette smoke exposure on skin barrier function and the rate of barrier function recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Suzaynn F Schick, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- Zuckerberg San Francisco General Hospital, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share the individual participant data (IPD) that underlie the results in our publications.
Supporting Information: Study Protocol
Time Frame: 9 months after publication
Access Criteria: Data will be made available to researchers who submit a detailed and well-supported description of their research plans.